CLINICAL TRIAL: NCT03438591
Title: The Effect of "Cerclage Pacing" for the Heart Failure Patients Who Need Cardiac Resynchronization Therapy (CRT): Early Feasibility Study
Brief Title: The Effect of "Cerclage Pacing" for the Heart Failure Patients Who Need Cardiac Resynchronization Therapy (CRT)
Acronym: Cerclage-CRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tau-MEDICAL Co., Ltd. (Industry)
Responsible Party: Principal Investigator, June-Hong Kim, MD, PhD, Professor, Pusan National University Yangsan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cerclage-CRT
Record Dates: First submitted 2018-02-13; First posted 2018-02-19 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Heart Failure; LBBB Complete
Keywords: cerclage pacing; cerclage-CRT; wide QRS
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: patients who meet the criteria of current CRT treatment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cerclage-CRT (medtronic 4196 lead) (Experimental): trans-coronary sinus intraseptal pacing (cerclage pacing) which technology to position the pacemaker lead into the septum for 'parahisian pacing'
  Interventions: Device: Medtronic 4196 lead

INTERVENTIONS:
Device: Medtronic 4196 lead — Cerclage-CRT pacing with Medtronic 4196 lead (Attain Ability Lead)

SUMMARY:
trans-coronary sinus intraseptal pacing (cerclage pacing)

DETAILED DESCRIPTION:
This study is aimed at looking at the effect of "Cerclage pacing" for the heart failure patients who need cardiac resynchronization therapy (CRT). The study hypothesis is that parahisian pacing by 'cerclage pacing' may have a similar benefit as is seen with permanent Hisian pacing

ELIGIBILITY:
Inclusion Criteria:

* who need cardiac resynchronization therapy (CRT) or CRT-non responder
* Left bundle branch block [LBBB]) > 120ms of QRS width
* Ejection fraction (EF) < 35%
* NYHA class III-IV in spite of optimal medical Tx

Exclusion Criteria:

* Unsuitable coronary vein anatomy on cardiac CT
* Subjects with prosthetic mechanical tricuspid valve
* Active infection
* Life expectancy less than 6 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
rate of procedural success | immediate postprocedure
  Narrowing QRS by 20% or greater compared with baseline QRS width

SECONDARY OUTCOMES:
Change in subjects' symptoms referred to NYHA Classification System | 12 months
  NYHA (New York Heart Association) : +1 grade
Change in subjects' improvement of parameters by Echocardiography | 12 months
  Ejection Fraction +5%
Change of Six minute walk Distance | 12 months
  improvement of SMWD
interrogation index of pacemaker lead | 12 months
  interrogation index of pacemaker lead

CONTACTS AND LOCATIONS:
Overall Officials: June-Hong Kim, MD, PhD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim JH, Hwang KW, Chon MK, Nam GB. Trans-coronary sinus intraseptal para-Hisian pacing: Cerclage pacing. Heart Rhythm. 2016 Apr;13(4):992-6. doi: 10.1016/j.hrthm.2015.12.002. Epub 2015 Dec 3. No abstract available. PMID 26654919